CLINICAL TRIAL: NCT05201378
Title: Deep Sclerectomy vs Xen in Solo Procedure: Comparative Study, Efficacy and Safety Profile
Brief Title: Deep Sclerectomy vs Xen in Solo Procedure
Acronym: SPXen
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SPXen
Record Dates: First submitted 2021-12-31; First posted 2022-01-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glaucoma is the leading cause of irreversible blindness in the world and the second leading cause of blindness after cataract after the age of 50. Lowering intraocular pressure (IOP) is the only treatment option to prevent visual field degradation. While medical treatment and selective laser trabeculoplasty are considered first-line options in open-angle glaucoma, the surgical option is considered in patients who have uncontrolled IOP under maximal tolerated medical treatment. In this situation, trabeculectomy or deep nonperforating sclerectomy may be performed. Although it is uncertain whether SPNP is superior to trabeculectomy, which is considered the gold standard of surgery, SPNP is a procedure that offers a better quality of life and fewer intra- and postoperative complications. SPNP was first described by Zimmerman. It consists in peeling off the internal wall of Schlemm's canal and the juxta-canalicular trabeculum which represent the main resistances to the evacuation of the aqueous humor. The trabecular meshwork is left intact and acts as a filter membrane between the subconjunctival space and the anterior chamber. The addition of mitomycin (MMC) is necessary because it is associated with better IOP control and greater surgical success. Although postoperative procedures such as needling or Nd:YAG laser-assisted gonioponctures are often required, SPNP offers good long-term results in patients who are naïve to any filtering surgery.

Minimally invasive surgery has been used more and more over the last 10 years. It aims to reduce surgical complications in comparison to classical filtering procedures while respecting the eye's own anatomy. Several devices have been invented to increase aqueous humor elimination. They can be implanted ab-interno or ab-externo and can be implanted in the suprachoroidal space, in Schlemm's canal or in the subconjunctival space. The XEN gelstent (Allergan, Dublin, Ireland) is placed ab-interno between the subconjunctival space and the anterior chamber, either in combination with cataract surgery or as a solo procedure.

The aim of the study is to compare the surgical success of these 2 techniques. No study has ever compared these 2 surgeries in solo procedure. A recent retrospective trial compared them in combined procedures without showing significant differences in IOP reduction. Nevertheless, the short follow-up period of 9 months may have been insufficient to show a real difference.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with primary or secondary open angle glaucoma
* Patient who has undergone a SPNP or XEN procedure in solo
* French speaking patient

Exclusion Criteria:

* Angle closure
* Less than 6 months follow-up
* History of eye filtering surgery included
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonperforating deep sclerectomy and XEN surgery patients in solo procedure between 01/01/2017 and 12/31/2018.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of surgical success at last visit in both groups | through study completion, an average of 6 months
  This outcome corresponds to intraocular pressure assessed at last visit, an average of 6 months.

SECONDARY OUTCOMES:
Intra- and postoperative complications | through study completion, an average of 6 months
  This outcome corresponds to the complications rate through study completion.
number of antiglaucoma medications | through study completion, an average of 6 months
  This outcome corresponds to the number of antiglaucoma medications at through study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Yves LACHKAR, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Causes of blindness and vision impairment in 2020 and trends over 30 years, and prevalence of avoidable blindness in relation to VISION 2020: the Right to Sight: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e144-e160. doi: 10.1016/S2214-109X(20)30489-7. Epub 2020 Dec 1. PMID 33275949
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Garg A, Vickerstaff V, Hunter R, Ambler G, Bunce C, Wormald R, Nathwani N, Barton K, Rubin G, Buszewicz M; LiGHT Trial Study Group. Selective laser trabeculoplasty versus eye drops for first-line treatment of ocular hypertension and glaucoma (LiGHT): a multicentre randomised controlled trial. Lancet. 2019 Apr 13;393(10180):1505-1516. doi: 10.1016/S0140-6736(18)32213-X. Epub 2019 Mar 9. PMID 30862377
- [Background] Eldaly MA, Bunce C, Elsheikha OZ, Wormald R. Non-penetrating filtration surgery versus trabeculectomy for open-angle glaucoma. Cochrane Database Syst Rev. 2014 Feb 15;2014(2):CD007059. doi: 10.1002/14651858.CD007059.pub2. PMID 24532137
- [Background] Rulli E, Biagioli E, Riva I, Gambirasio G, De Simone I, Floriani I, Quaranta L. Efficacy and safety of trabeculectomy vs nonpenetrating surgical procedures: a systematic review and meta-analysis. JAMA Ophthalmol. 2013 Dec;131(12):1573-82. doi: 10.1001/jamaophthalmol.2013.5059. PMID 24158640
- [Result] Touboul A, Fels A, Morin A, Bensmail D, Lachkar Y. One-Year Outcomes of Standalone XEN Gel Stent Versus Nonpenetrating Deep Sclerectomy. J Glaucoma. 2022 Dec 1;31(12):955-965. doi: 10.1097/IJG.0000000000002108. Epub 2022 Aug 22. PMID 36001498